CLINICAL TRIAL: NCT00705926
Title: A Phase 1 Clinical Trial to Evaluate the Initiation of Treatment Versus no Treatment During Acute HIV-1 Infection
Brief Title: Effectiveness of Antiretroviral Therapy During Acute HIV Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Eric Rosenberg, MD, Investigator of Record, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AI071915 (NIH); RO1AIO71915 (Other Grant/Funding Number: NIAID)
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: HIV Infections
Keywords: Acute Infection; HIV; HAART; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Antiretroviral Therapy, Highly Active

ARMS (3):
- A1 (Experimental): Antiretroviral therapy followed by discontinuation at Week 12.
  Interventions: Drug: Highly Active Antiretroviral Therapy (HAART)
- A2 (Experimental): Antiretroviral therapy followed by discontinuation at Week 32.
  Interventions: Drug: Highly Active Antiretroviral Therapy (HAART)
- B (Placebo Comparator): No treatment.
  Interventions: Other: No treatment

INTERVENTIONS:
Drug: Highly Active Antiretroviral Therapy (HAART) — Participants in Groups A1 and A2 will receive HAART for either 12 or 32 weeks. Their medications will not be provided by the study.
  Arms: A1; A2
Other: No treatment — Participants in this group will not receive treatment at this stage of their infection.
  Arms: B

SUMMARY:
This study will determine whether HIV treatment that is initiated during the acute phase of HIV infection, followed by discontinuation of treatment, is effective in reducing the amount of HIV and an increasing the amount of CD4 cells in the blood of people with HIV, compared to the amounts of HIV and CD4 cells in people who do not receive treatment at this stage.

DETAILED DESCRIPTION:
Antiretroviral (ARV) therapy for the treatment of HIV infection has been remarkably successful in reducing morbidity and mortality in HIV infected people. This treatment still has its shortcomings, however. Individuals receiving ARV treatment are at risk of toxicity, developing drug resistance, and unknown long-term side effects. Therefore, development of alternative treatment strategies is important. A short course of ARV treatment that is initiated during the acute period of HIV infection, followed by treatment cessation may have a substantial impact on controlling infection and delaying the need for lifelong potent ARV therapy. The purpose of this study is to investigate whether treatment initiated during acute HIV infection and followed by a terminal treatment interruption is effective in lowering the viral load set point and raising CD4 cell counts in people with HIV, as compared to those measures in people with HIV who have received no treatment.

Participants in this study will be randomly assigned to one of three groups. Participants in Group A1 will receive ARV therapy for 12 weeks. Participants in Group A2 will receive ARV therapy for 32 weeks. Participants in Group B will not receive any treatment. This study will not provide medications to any of the groups. All groups will be followed for a total of 72 weeks following study entry. Participants will attend between 30 and 36 study visits over the course of the 72 weeks, depending on their study group. Study visits will occur every week for the first 12 weeks and then every 1 to 6 weeks for the remainder of the study. Tests occurring at study visits may include blood tests, investigational immune system tests, and pregnancy tests. Participants will also undergo a complete physical exam and will be asked to provide information about their medical and medication histories.

ELIGIBILITY:
Inclusion Criteria:

* Acute HIV infection as determined by a positive HIV viral load (at least 5,000 copies of RNA per ml of plasma) and a negative or indeterminate Western Blot test
* Certain laboratory values. More information about this criterion can be found in the protocol.
* Agrees to use an approved form of contraception

Exclusion Criteria:

* Presence of opportunistic infections or AIDS-defining illnesses, unless they are directly attributable to the acute seroconversion illness
* Receipt of investigational research agents within 30 days prior to study entry
* Receipt of prior experimental HIV vaccines. Individuals who received a saline placebo in a prior HIV vaccine trial are not excluded, provided that they did not receive a sham vector or an adjuvant.
* Receipt of immunosuppressive medications or immunomodulators (e.g., cytokine therapy) within the past 6 months. Participants taking corticosteroid nasal spray for allergic rhinitis; topical corticosteroids for acute, uncomplicated dermatitis; or over the counter medications for acute, uncomplicated dermatitis for a period not longer than 14 days will not be excluded.
* Current use of prohibited concomitant medications
* Current anti-tuberculosis prophylaxis or therapy
* Serious illness other than acute HIV infection requiring systemic treatment or hospitalization until either therapy is completed or patient is clinically stable on therapy
* Hepatitis B surface antigen positivity within 21 days prior to study entry
* Pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-10; Primary Completion 2013-02-07 (Actual); Study Completion 2017-07-16 (Actual)

PRIMARY OUTCOMES:
Difference in the level of HIV RNA at viral load set point if therapy is initiated during acute HIV infection followed by terminal treatment interruption after 12 or 32 weeks of treatment compared to that under no treatment | Week 72

SECONDARY OUTCOMES:
Difference in the level of CD4 cells if therapy is initiated during acute HIV infection followed by terminal treatment interruption after 12 or 32 weeks of treatment compared to that under no treatment | Week 72
Difference in the level of HIV RNA and CD4 cell numbers between therapy initiated during acute HIV infection followed by terminal treatment interruption after at least 12 weeks of treatment and no therapy at 16 weeks after discontinuation of treatment | Weeks 12 and 16
Difference in the level of HIV at viral load set point and CD4 cell number at 72 weeks after study entry if therapy is initiated during acute HIV infection followed by terminal treatment interruption at 12 weeks versus at 32 weeks | Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Eric S. Rosenberg, MD, Study Chair — Massachusetts General Hospital, Division of Infectious Diseases; H.T. Banks, PhD, Principal Investigator — North Carolina State University, College of Physical and Mathematical Sciences; Marie Davidian, PhD, Principal Investigator — North Carolina State University, Department of Statistics
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Kassutto S, Maghsoudi K, Johnston MN, Robbins GK, Burgett NC, Sax PE, Cohen D, Pae E, Davis B, Zachary K, Basgoz N, D'agata EM, DeGruttola V, Walker BD, Rosenberg ES. Longitudinal analysis of clinical markers following antiretroviral therapy initiated during acute or early HIV type 1 infection. Clin Infect Dis. 2006 Apr 1;42(7):1024-31. doi: 10.1086/500410. Epub 2006 Feb 27. PMID 16511771
- [Background] Kassutto S, Rosenberg ES. Editorial comment: treatment of acute HIV infection--uncertainties about best practice. AIDS Read. 2005 May;15(5):250-1. No abstract available. PMID 15900635
- [Background] Kassutto S, Rosenberg ES. Primary HIV type 1 infection. Clin Infect Dis. 2004 May 15;38(10):1447-53. doi: 10.1086/420745. Epub 2004 Apr 30. PMID 15156484
- [Background] Lacabaratz-Porret C, Urrutia A, Doisne JM, Goujard C, Deveau C, Dalod M, Meyer L, Rouzioux C, Delfraissy JF, Venet A, Sinet M. Impact of antiretroviral therapy and changes in virus load on human immunodeficiency virus (HIV)-specific T cell responses in primary HIV infection. J Infect Dis. 2003 Mar 1;187(5):748-57. doi: 10.1086/368333. Epub 2003 Feb 18. PMID 12599048
- [Background] Malhotra U, Berrey MM, Huang Y, Markee J, Brown DJ, Ap S, Musey L, Schacker T, Corey L, McElrath MJ. Effect of combination antiretroviral therapy on T-cell immunity in acute human immunodeficiency virus type 1 infection. J Infect Dis. 2000 Jan;181(1):121-31. doi: 10.1086/315202. PMID 10608758